CLINICAL TRIAL: NCT06530823
Title: Pemigatinib Combined With Durvalumab for the Safety and Efficacy in Second-Line Treatment of Biliary Tract Cancer: A Single-Arm, Multicenter Phase II Clinical Trial
Brief Title: Pemigatinib Combined With Durvalumab for Previously Treated Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Chairman of Clinical Research Institute, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2024-H018-P001
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Biliary Tract Carcinoma; Cholangiocarcinoma
Keywords: biliary tract carcinoma; cholangiocarcinoma; FGFR mutation; targeted thearpy; immunotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pemigatinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pemigatinib and Durvalumab (Experimental): The combination of targeted drugs and immunotherapies has demonstrated their clinical value in the treatment of various tumors, and pemigatinib and durvalumab are such a promising combination product. In this combination, Pemigatinib is used according to the following rules:13.5mg, oral administration, once daily, swallow the entire tablet with or without food. Take for 2 weeks and then discontinue for 1 week.
  Durvalumab is used as this: 1500mg, intravenous infusion, once every three weeks. Each infusion should take over 60 minutes.
  Interventions: Drug: Pemigatinib and Durvalumab

INTERVENTIONS:
Drug: Pemigatinib and Durvalumab — Pemigatinib combined with Durvalumab Pemigatinib: 13.5mg, oral administration, once daily, swallow the entire tablet with or without food. Take for 2 weeks and then discontinue for 1 week. Durvalumab: 1500mg, intravenous infusion, once every three weeks. Each infusion should take over 60 minutes.

SUMMARY:
This study is a single-arm, multicenter Phase II clinical trial designed to preliminarily assess the safety and efficacy of the combination therapy of pemigatinib and durvalumab in the second-line treatment of patients with advanced malignant biliary tract cancer.

The study anticipates enrolling 38 participants characterized by the following criteria: 1) A confirmed diagnosis of advanced, metastatic, or unresectable biliary tract cancer by histopathological examination; 2) Presence of FGFR2 fusion or rearrangement confirmed by testing; 3) Prior receipt of first-line treatment for biliary tract cancer.

The primary questions the study aims to address are:

1. Can the combination of pemigatinib and durvalumab improve the prognosis of participants with previously treated biliary tract cancer (BTC)?
2. What is the safety profile of the treatment with pemigatinib and durvalumab?

Participants will receive:

1. Oral administration of 13.5 mg pemigatinib once daily, in combination with durvalumab 1500 mg via intravenous infusion.
2. Follow-up visits will be scheduled every 6 weeks.

Investigators will observe and document the objective tumor response rate of the participants, as well as progression-free survival (PFS), disease control rate (DCR), overall survival (OS), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, men and women;
2. ECOG performance status of 0-1;
3. Histologically confirmed advanced gallbladder cancer or cholangiocarcinoma patients who have received one prior line of therapy;
4. Adult patients with advanced, metastatic, or unresectable cholangiocarcinoma or gallbladder cancer confirmed to have FGFR2 fusion or rearrangement;
5. Diagnosed with locally advanced disease according to the 8th edition of AJCC, with clinical staging of cT3/4NxM0/1 for gallbladder cancer, intrahepatic cholangiocarcinoma, or hilar cholangiocarcinoma, or cT2N2M0, cT3/4NxM0/1 for distal cholangiocarcinoma based on enhanced CT or MRI;
6. Use of contraception during the study period;
7. Life expectancy ≥3 months;
8. All patients must provide tumor tissue specimens (fresh or paraffin-embedded) for FGFR2 expression analysis before enrollment and after surgery (5 slides within 3 years are required);
9. At least one measurable lesion according to RECIST 1.1 criteria, which has not been irradiated;
10. Within 7 days prior to the first administration of the study drug, the organ function levels of the enrolled patients must meet the following requirements:

    1. Hematopoietic function: Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count (PLT) ≥ 100×10^9/L, hemoglobin (Hb) ≥90g/L, and no blood transfusion or component blood transfusion within 14 days prior to testing;
    2. Hepatic function: Serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (APK) ≤2.5 times ULN, serum creatinine ≤1.5 times ULN and creatinine clearance (based on the Cockcroft-Gault formula) ≥50mL/min, serum albumin (ALB) ≥30g/L, Child-Pugh class A;
    3. Coagulation function: For patients not receiving anticoagulant therapy, international normalized ratio (INR), activated partial thromboplastin time (APTT) ≤1.5 times ULN; patients receiving anticoagulant therapy should maintain therapeutic levels of anticoagulants;
    4. Thyroid function: Thyroid-stimulating hormone (TSH) ≤1×ULN, if TSH >1×ULN, free T3 (FT3) and free T4 (FT4) levels should also be assessed, and if normal, the patient may be enrolled;
    5. Renal function: Urine protein ≤1+. If urine protein >1+, a 24-hour urine protein test is required, and the total amount must be ≤1 gram for enrollment;
    6. Normal cardiac function, i.e., normal electrocardiogram or clinically insignificant abnormalities, and left ventricular ejection fraction (LVEF) >50% as shown by echocardiography;
11. Serum pregnancy test results must be negative within 7 days prior to the first administration of the trial medication for women of childbearing age; men with reproductive capacity or women who may become pregnant must use highly effective contraception (e.g., oral contraceptives, intrauterine devices, abstinence, or barrier methods combined with spermicides) throughout the trial and continue for 12 months after treatment;
12. Volunteers willing to participate in the study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Patients who have not received standard first-line treatment for advanced biliary tract tumors;
2. Pregnant or breastfeeding women, and women of childbearing age with positive pregnancy test results at baseline;
3. Patients diagnosed with central nervous system metastasis by CT/MR/PET-CT;
4. Patients who have previously received live vaccine administration or other antitumor treatments such as radiotherapy;
5. Patients who have participated in or are currently participating in other drug or therapy clinical trials within 4 weeks prior to the first administration of the study medication;
6. Patients who have undergone major surgical procedures within 4 weeks prior to the first administration of the study medication or have not recovered from the side effects of such surgery, or patients who have undergone radiotherapy within 2 weeks prior to the first administration of the study medication;
7. Patients with any primary immunodeficiency, active autoimmune disease, or history of autoimmune disease, including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, vitiligo, patients with a history of asthma who have completely resolved in childhood and do not require any intervention in adulthood may be included; patients with asthma requiring medical intervention with bronchodilators are excluded;
8. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation, and patients currently using immunosuppressants or corticosteroids for immunosuppressive purposes (dosage >10mg/day prednisone or other equivalent corticosteroids) and still in use within 2 weeks prior to enrollment;
9. Patients with other malignancies within the past 5 years, except for cured skin basal cell or squamous cell carcinoma, superficial bladder cancer, early prostate cancer, in situ cervical cancer, or breast cancer;
10. Patients who have received hematopoietic growth factors within 1 week prior to the first administration of the study medication, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc.;
11. Patients with positive HIV antibodies or syphilis antibodies, and patients with active hepatitis B or C;
12. Known allergies to recombinant humanized PD-L1 monoclonal antibody drugs and their components;
13. Patients with symptomatic pleural effusion, pericardial effusion, or ascites requiring clinical treatment;
14. Patients with severe cardiovascular diseases within the last 12 months, such as clinically significant coronary heart disease, NYHA≥II congestive heart failure, uncontrolled arrhythmias, myocardial infarction;
15. Within 6 months prior to the first administration of the study medication, the following conditions have occurred: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmias or angina; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism.
16. Patients who have undergone any type of gastrointestinal surgery, or have upper gastrointestinal obstruction, bleeding, digestive dysfunction, or malabsorption syndrome that may affect the absorption of the study medication;
17. Concurrent severe uncontrollable infections or other severe uncontrollable comorbidities, moderate or severe renal impairment;
18. Active pulmonary diseases, such as interstitial pneumonia, pneumonia, chronic obstructive pulmonary disease, asthma, or a history of active tuberculosis.
19. Abnormal coagulation function (INR>2.0, PT>16s), with a tendency to bleed or currently receiving thrombolytic or anticoagulant therapy, prophylactic use of low-dose aspirin, low molecular weight heparin is allowed;
20. Significant clinical bleeding symptoms or a clear tendency to bleed within 3 months, such as coughing or expectorating blood ≥2.5ml, history of gastrointestinal bleeding, esophageal and gastric varices with bleeding risk, bleeding gastric ulcers or patients with vasculitis, etc.; if the baseline fecal occult blood test is positive, it can be retested, and if it is still positive after retesting, a gastroscopy is required, and if gastroscopy indicates severe esophageal and gastric varices, the patient may not be enrolled (patients who have undergone gastroscopy within 3 months and excluded such conditions are excluded);
21. Known genetic or acquired bleeding and thrombotic tendencies, such as hemophilia, coagulation disorders, thrombocytopenia, etc.;
22. History of substance abuse that cannot be quit or history of mental disorders.
23. Use of warfarin or any other coumarin derivative anticoagulants within 14 days prior to the first administration of the study medication.
24. Other severe, acute, or chronic medical diseases or laboratory abnormalities that the investigator judges may increase the risk associated with participating in the study or may interfere with the interpretation of the study results.
25. Patients deemed to have poor compliance by the investigator, or other conditions that make them unsuitable for participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From enrollment to the end of treatment at 8 weeks
  Objective response rate is defined as the proportion of subjects who achieved a complete response (CR; disappearance of all target lesions) or a PR (> 30% decrease in the sum of the longest diameters of target lesions) based on RECIST v1.1. Clinical response will be determined by an independent radiological review committee.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS=first dose to progression disease [PD] or death
Disease Control Rate (DCR) | From enrollment to the end of treatment at 8 weeks
  DCR=CR+PR+satble disease
Overall survival (OS) | From date of randomization until the date of death from any cause, whichever came first, assessed up to 36 months
  OS=first dose to death of any cause
Adverse Event (AE) | From enrollment to the end of treatment at 8 weeks

IPD SHARING:
Plan to Share IPD: No